CLINICAL TRIAL: NCT02844400
Title: Assessing Performance Status in Cancer Patients Using Cardiopulmonary Exercise Testing and Wearable Data Generation: A Prospective Observational Study
Brief Title: Cancer Patients' Performance Status Assessed Using Cardiopulmonary Exercise Testing and Wearable Data Generation
Status: Completed | Type: Observational
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: LCCC 1605
Record Dates: First submitted 2016-07-21; First posted 2016-07-26 (Estimated); Last update posted 2019-02-22 (Actual); Status verified 2019-02

CONDITIONS: Malignant Solid Tumor; Hematologic Malignancies
MeSH Terms: conditions — Hematologic Neoplasms | interventions — Exercise Test

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Adjuvant and Curative Chemotherapy: 30 participants. Primarily older (60+ years in age) cancer patients receiving cytotoxic chemotherapy with adjuvant or curative intent. Will undergo both the Physical Performance Testing and Biometric Devices interventions.
  Interventions: Device: Biometric Devices; Other: Physical Performance Testing
- Palliative Chemoteraphy: 30 participants. Primarily older (60+ years in age) cancer patients receiving cytotoxic chemotherapy with palliative intent. Will undergo both the Physical Performance Testing and Biometric Devices interventions.
  Interventions: Device: Biometric Devices; Other: Physical Performance Testing

INTERVENTIONS:
Device: Biometric Devices — Patients will wear two devices: HealthPatch Sensor and Phillips Actiwatch. Health data (e.g. average steps per day, resting heart rate) will be collected and monitored over the course of a cycle of cytotoxic chemotherapy.
Other: Physical Performance Testing — Patients will complete a CPET and 6 minute walk test within one week of starting an upcoming chemotherapy cycle and they will undergo a second CPET upon completion of said chemotherapy cycle.

SUMMARY:
The primary objective of this study is to establish the feasibility and value of physical fitness assessment within patients receiving cytotoxic chemotherapy. If successful, this project will establish the groundwork for physical function assessment in larger cancer clinical trials to assist patient selection and evaluation of toxicity and/or response among trial participants.

DETAILED DESCRIPTION:
Physical fitness, whether measured by performance capacity or daily activity, can predict risk of toxicity while helping to evaluate toxicity itself in the course of cancer chemotherapy. Cytotoxic chemotherapy causes premature aging and frailty in many cancer patients, so measuring and improving physical function may also limit late morbidity and mortality. Clinician-rated performance status (cPS; e.g., ECOG or Karnofsky PS) with or without concomitant organ function testing is the usual gold standard for risk prognostication and patient selection in most cancer settings, but cPS is subjective, unreliable, and relatively sensitive only for patients with significant functional compromise. Objective evaluations of physical function have the potential to augment or even replace cPS in the cancer treatment setting.

ELIGIBILITY:
Inclusion Criteria:

* Patients receiving cytotoxic chemotherapy with at least a 3 week cycle (either adjuvant/curative or palliative)
* Age ≥ 18, prioritizing patients ≥ 60 years
* At least 6 weeks out from surgical resection
* Presence of working email address
* Access to internet at home and either access to wireless internet or cellular data reception
* Ability to read and understand English
* Ability to understand and comply with study procedures

Exclusion Criteria:

* Dementia, altered mental status, or psychiatric condition that would prohibit the understanding or rendering of informed consent
* Contraindication to CPET per standard American Thoracic Society (ATS) guidelines

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 60 patients with cancer undergoing a cycle of cytotoxic chemotherapy.
Sampling Method: Non-Probability Sample
Enrollment: 67 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Proportion of patients being approached that agree to participate in the study | 12 months
  Measure 1 for study feasibility
Proportion of patients who complete both baseline and follow up CPET tests without significant testing-related adverse events | 12 months
  Measure 2 for study feasibility
Proportion of patients who wear HealthPatch and have data captured successfully for at least 75% of the time | 12 months
  Measure 3 for study feasibility
Patients who wear Philips Actiwatch and have data captured successfully for at least 75% of the time | 12 months
  Measure 4 for study feasibility
Proportion of patients for whom all data is successfully recorded within the database | 12 months
  Measure 5 for study feasibility

SECONDARY OUTCOMES:
VO2max measured both pre- and post-chemotherapy | 12 months
  Measured via cycle egometry
6 Minute Walk Distance (6MWD) | 12 months
Patient-reported sympotomatic toxicity and quality of life | 12 months
  Measured using PROMIS, PRO-CTCAE, Godin Leisure Time Exercise questionnaires and Geriatric Assessment
Patient activity/steps per day | 12 months
  Measured using Philips Actiwatch
Heart rate | 12 months
  Continuous heart rate data, resting heart rate, and heart rate variability will be measured using HealthPatch
Clinician-rated performance status | 12 months
  Clinician-rated ECOG and Karnofsky Performance Status (KPS)
Incidence and number of falls | 12 months
  Measured by HealthPatch
Sleep duration | 12 months
  Measured by Philips Actiwatch

CONTACTS AND LOCATIONS:
Overall Officials: Natalie Grover, MD, Principal Investigator — University of North Carolina, Chapel Hill; William A Wood, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: UNC Lineberger Comprehensive Cancer Center — http://unclineberger.org